CLINICAL TRIAL: NCT03059004
Title: Treatment of Meniscal Problems in Osteoarthritis
Brief Title: Comparing Different Types of Physical Therapy for Treating People With a Meniscal Tear and Osteoarthritis
Acronym: TeMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); State University of New York at Buffalo (Other); The Cleveland Clinic (Other); University of Pittsburgh (Other); University of Melbourne (Other); Boston University (Other)
Responsible Party: Principal Investigator, Jeffrey Neil Katz, MD, Associate Physician, Brigham and Women's Hospital Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01AR071658-01 (NIH)
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Meniscal Degeneration; Osteoarthritis, Knee
Keywords: physical therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Four arm parallel randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will not be appraised of treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. Home Exercise Program (Experimental): The Home Exercise group receives the TeMPO Home Exercise Program (including a set of weights, a DVD showing how to complete the TeMPO exercises, and a pamphlet outlining instructions on how to complete the exercises and how often should they be done).
  Interventions: Behavioral: TeMPO Home Exercise Program
- 2. Home Exercise Program + SMS Messages (Experimental): Subjects in this arm receive the TeMPO Home Exercise Program and motivational SMS messages to encourage them to adhere to the TeMPO Home Exercise regimen.
  Interventions: Behavioral: TeMPO Home Exercise Program; Behavioral: Motivational SMS Messages
- 3. In-Clinic Topical Therapy (Experimental): Subjects in this arm receive the TeMPO Home Exercise Program, motivational SMS messages to encourage them to adhere to the TeMPO Home Exercise Program, and 14 in-clinic sessions with a trained physical therapist. The therapist will apply topical therapies: ultrasound, gel, and manual therapy.
  Interventions: Behavioral: TeMPO Home Exercise Program; Behavioral: Motivational SMS Messages; Behavioral: In-Clinic Topical Therapy
- 4. In-Clinic Exercise Therapy (Experimental): Subjects in this arm will receive the TeMPO Home Exercise Program, SMS motivational messages to encourage them to adhere to the TeMPO Home Exercise Program and 14 in-clinic sessions with a trained physical therapist. The therapist will supervise the participant in a rigorous set of strengthening and stretching exercises.
  Interventions: Behavioral: TeMPO Home Exercise Program; Behavioral: Motivational SMS Messages; Behavioral: In-Clinic Exercise Therapy

INTERVENTIONS:
Behavioral: TeMPO Home Exercise Program — This exercise program includes quadriceps, gluteus medius, gluteus maximus, and core exercises. The program includes a DVD and multi-page instruction pamphlet.
Behavioral: Motivational SMS Messages — The motivational SMS messages will be sent three times per week encouraging participants to complete their exercises.
  Arms: 2. Home Exercise Program + SMS Messages; 3. In-Clinic Topical Therapy; 4. In-Clinic Exercise Therapy
Behavioral: In-Clinic Topical Therapy — Subjects will be assigned to a physical therapist and will attend 14 in-clinic topical therapy sessions. Sessions will include application of ultrasound, gel, and manual therapy.
  Arms: 3. In-Clinic Topical Therapy
Behavioral: In-Clinic Exercise Therapy — Subjects will be assigned to a physical therapist and will attend 14 in-clinic exercise and manual therapy sessions. Sessions will include the same exercises from the Home Exercise Program but the in-clinic therapy setting will allow for more personalization.
  Arms: 4. In-Clinic Exercise Therapy

SUMMARY:
Knee osteoarthritis is a disabling problem affecting over 15 million adults in the United States. Many people who have knee arthritis also experience painful meniscal tears. There are a number of different treatments that can be used to manage meniscal tears in the presence of knee arthritis. Treatments include surgically removing the damaged part of the meniscus; strengthening exercises to improve pain and function; manual therapy including massage and mobilization; acupuncture; and others. The combination of surgery and exercise therapy was long thought to be the best treatment. However, recent studies have shown that surgery followed by physical therapy is no more effective than physical therapy by itself.

While physical therapy alone has been shown to result in similar pain relief as arthroscopic surgery, researchers have not yet done studies to determine what type of physical therapy is best for people with knee arthritis and meniscal tears. In the "TeMPO" Trial, we will be comparing 4 different, non-operative physical therapy regimens in order to gain a better understanding of how physical therapy works and what regimen will best reduce pain and improve function in persons with meniscal tear and osteoarthritis. The four arms in this randomized trial will contain different combinations of therapeutic treatments including in-clinic therapist-supervised exercise, in-clinic topical therapies, and exercises to be completed at home. Subjects in three of the arms will also receive motivational SMS (text) messages intended to improve adherence to the home exercise regimen.

TeMPO is designed as a randomized controlled trial. Participants will be assigned randomly to one of the four arms. All arms include therapies that have been previously shown to work in clinical settings. One arm also contains some placebo treatments. The placebo treatments will help us to understand what aspects of physical therapy actually make people feel better.

Our hypothesis is that subjects in the arm that includes in-clinic physical therapy and a home exercise regimen will experience more pain relief than subjects in each of the other arms. Also, we expect that subjects in the arm that receives the home exercise regimen and SMS messages will experience more pain relief than subjects in the arm that receives home exercise without the SMS messages.

DETAILED DESCRIPTION:
Knee osteoarthritis is a disabling problem affecting over 15 million adults in the United States. Many people who have knee arthritis also experience painful meniscal tears. There are a number of different treatments that can be used to address meniscal tears in the presence of knee arthritis. These include surgically removing the damaged part of the meniscus; strengthening exercises; manual therapy including massage and mobilization; and others. The combination of surgery and exercise therapy was long thought to be the best treatment. However, recent studies have shown that surgery followed by physical therapy leads to similar levels of pain relief as physical therapy alone.

While physical therapy appears to be useful in knee osteoarthritis and meniscal tear, research is needed to determine what type of physical therapy is best for people with these conditions. The "TeMPO" Trial will compare 4 different non-operative regimens in order to gain a better understanding of how physical therapy works and to determine which regimen will best reduce participants' pain and improve their function. The four arms in this trial will contain different combinations of therapeutic treatments including in-clinic supervised exercise therapy, in-clinic topical therapies, and exercises to be completed at home. Some of the arms will also receive text messages designed to improve adherence to assigned exercises. All arms include therapies that have been previously shown to work in clinical settings. One arm also contains some placebo treatments. The placebo treatments will help identify the aspects of physical therapy that make people feel better.

The four arms in the TeMPO study are as follows:

1. Home Exercise Program
2. Home Exercise Program + Motivational SMS messages
3. Home Exercise Program + Motivational SMS messages + In-Clinic topical therapy
4. Home Exercise Program + Motivational SMS messages + In-Clinic Exercise Therapy

ELIGIBILITY:
Inclusion Criteria:

* Knee pain of at least 21 days duration if traumatic; no minimum duration if non-traumatic
* Age 45 -85 years
* Physician diagnosis of meniscal tear
* Evidence on MRI of meniscal tear
* Evidence of osteoarthritic changes on imaging: Cartilage damage on MRI, osteophyte or joint space narrowing on X-ray

Exclusion Criteria:

* KL-Grade 4
* Inflammatory arthritis
* Prior APM or TKR on index knee; or any surgery on index knee in prior 6 mo
* Pregnancy
* Contraindication to MRI
* Daily use of strong opioids
* Intra-articular therapy in last 4 weeks
* Non-English speaking
* History of dementia
* Currently resides in a nursing home
* Current claimant of worker's compensation for this condition

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 879 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Randomization to 3 months
  Difference between arms in change in the KOOS Pain score over three months (Arm 4 vs. Arm 1; Arm 4 vs. Arm 2; Arm 2 vs. Arm 1. Arm 4 vs. Arm 3)

SECONDARY OUTCOMES:
Change in function | Randomization to 3 months
  Difference between arms in change in the KOOS ADL score over three months (Arm 4 vs. Arm 1; Arm 4 vs. Arm 2; Arm 2 vs. Arm 1; Arm 4 vs. Arm 3)
Change in quality of life | Randomization to 3 months
  Difference between arms in change in quality of life measured with the EQ-5D scale over three months (Arm 4 vs. Arm 1; Arm 4 vs. Arm 2; Arm 2 vs. Arm 1; Arm 4 vs. Arm 3)
Binary treatment failure indicator | Randomization to 3 months
  Difference between arms in treatment failure defined as either not reaching improvement of >=8 points on KOOS Pain or receiving injection or undergoing index knee surgery within three months (Arm 4 vs. Arm 1; Arm 4 vs. Arm 2; Arm 2 vs. Arm 1; Arm 4 vs. Arm 3)
Forty meter fast-paced walk | Randomization to 3 months
  Difference between arms in change in 40 m fast-paced walk (seconds) over three months (Arm 4 vs. Arm 1; Arm 4 vs. Arm 2; Arm 2 vs. Arm 1; Arm 4 vs. Arm 3)
30-second sit to stand | Randomization to 3 months
  Difference between arms in number of repetitions (of sit to stand) over 30 seconds
Strength of quadriceps, hamstrings, gluteus medius | Baseline to 3 months
  Difference between arms in strength (pounds-cm) between arms, measured at three sites (quadriceps, hamstrings, gluteus medius)
Single Leg Balance | Baseline to 3 months
  Difference between arms in number of seconds participant can stand on single leg without moving hands off hips, stepping or stumbling, abducting or flexing hip beyond 30 deg, lifting heel or forefoot off ground.
Durability of pain relief | 3-12 months
  Difference between arms in proportion of subjects who maintain through 12 months the benefit (in KOOS Pain) achieved at 3 months. (Arm 4 vs. Arm 1; Arm 4 vs. Arm 2; Arm 2 vs. Arm 1; Arm 4 vs. Arm 3 )

CONTACTS AND LOCATIONS:
Overall Officials: Chuck Washabaugh, PhD, Study Chair — National Institute for Arthritis, Musculoskeletal and Skin Diseases (NIAMS, NIH)
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University at Buffalo Medical Department, Buffalo, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Upon request to jnkatz@bwh.harvard.edu we will share core baseline and primary outcome data 12 months after primary report is published. Request must include hypotheses, analytic plans, rationale.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 12 months after publication of primary trial manuscript
Access Criteria: note to PI, jnkatz@bwh.harvard.edu with rationale, significance analysis plan.

REFERENCES:
- [Derived] Katz JN, Collins JE, Bisson L, Jones MH, Irrgang JJ, Selzer F, Safran-Norton CE, Spindler KP, Yang HY, Shrestha S, Bennell KL, Sullivan JK, Kluczynski MA, Arant K, Opare-Addo M, Huizinga JL, Zimmerman Z, Sople D, Tonsoline P, Kale M, Wind WM Jr, Chen AF, Freitas M, Lesniak B, Jordan K, Matzkin EG, Dawson C, Farrow L, Musahl V, Leddy JJ, Martin SD, Losina E. A Randomized Trial of Physical Therapy for Meniscal Tear and Knee Pain. N Engl J Med. 2025 Oct 30;393(17):1694-1703. doi: 10.1056/NEJMoa2503385. PMID 41160820
- [Derived] Safran-Norton CE, Sullivan JK, Irrgang JJ, Kerman HM, Bennell KL, Calabrese G, Dechaves L, Deluca B, Gil AB, Kale M, Luc-Harkey B, Selzer F, Sople D, Tonsoline P, Losina E, Katz JN. A consensus-based process identifying physical therapy and exercise treatments for patients with degenerative meniscal tears and knee OA: the TeMPO physical therapy interventions and home exercise program. BMC Musculoskelet Disord. 2019 Nov 4;20(1):514. doi: 10.1186/s12891-019-2872-x. PMID 31684921
- [Derived] Sullivan JK, Irrgang JJ, Losina E, Safran-Norton C, Collins J, Shrestha S, Selzer F, Bennell K, Bisson L, Chen AT, Dawson CK, Gil AB, Jones MH, Kluczynski MA, Lafferty K, Lange J, Lape EC, Leddy J, Mares AV, Spindler K, Turczyk J, Katz JN. The TeMPO trial (treatment of meniscal tears in osteoarthritis): rationale and design features for a four arm randomized controlled clinical trial. BMC Musculoskelet Disord. 2018 Dec 1;19(1):429. doi: 10.1186/s12891-018-2327-9. PMID 30501629

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT03059004/SAP_000.pdf